CLINICAL TRIAL: NCT07096115
Title: The 90% Effective Dose of Taiglididine for Inhibiting Laryngeal Mask Insertion Response in Elderly Patients
Brief Title: ED90 of Teglidine for Suppressing LMA Insertion Response in the Elderly
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First People's Hospital of Lianyungang (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KY-20250324002-01
Record Dates: First submitted 2025-06-26; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Urological Surgery
Keywords: Taiglididine; Elderly Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Taiglididine Sequential Dose-Finding for LMA Insertion Suppression (Experimental)
  Interventions: Drug: Taiglididine

INTERVENTIONS:
Drug: Taiglididine — The first patient receives an intravenous injection of 1 mg taiglididine for anesthesia induction, followed by 1-2 mg/kg propofol. When the patient's bispectral index (BIS) drops below 60, eyelash reflex disappears, and MOAA/S score is 0, intravenous rocuronium 0.6 mg/kg is given, and a laryngeal mask is inserted by a senior anesthesiologist using a unified method 1 min later. From the second patient onward, the taiglididine dose is dynamically adjusted based on the previous patient's response to laryngeal mask insertion using BCD-UDM: if the previous patient shows a positive insertion response (positive response or MOAA/S ≥2 within 2 min after induction), the next patient's dose increases by 0.1 mg; if negative, a random number (1-95) generated by computer determines the dose: doses remain unchanged when the number is 6-95 (89% probability) and decrease by 0.1 mg when the number is 1-5 (11% probability). A collaborator not involved in result evaluation provides a sealed envelope with

SUMMARY:
This research protocol aims to investigate the 90% effective dose (ED90) of taiglididine for inhibiting laryngeal mask insertion response in elderly patients. It is a non-randomized controlled trial using a biased coin design up-down method (BCD-UDM). A total of 54 elderly patients aged 65-80 years with ASA I-III, BMI 18-30 kg/m², and suitable for urological surgery under general anesthesia with laryngeal mask insertion will be enrolled. The first patient receives an intravenous injection of 1 mg taiglididine, followed by propofol and rocuronium. Subsequent doses of taiglididine are adjusted dynamically based on the previous patient's response: increasing by 0.1 mg if the insertion response is positive, or using BCD-UDM (11% probability to decrease by 0.1 mg, 89% to remain) if negative. The primary efficacy endpoint is the occurrence of laryngeal mask insertion response, while secondary endpoints include adverse events, vital sign changes, insertion success rate, and various time intervals. Safety is evaluated by monitoring vital signs. Statistical analysis will use SPSS 25.0 and R software to calculate ED90 and 95% confidence intervals via probit regression and bootstrap method, with at least 45 valid patients required to complete the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 65-80 years old.
2. ASA physical status I-III.
3. BMI 18-30 kg/m² (inclusive of critical values).
4. Mallampati class I or II, mouth opening >2.5 cm.
5. No abnormal airway or head/neck conditions.
6. No risk of reflux or aspiration (e.g., full stomach, obesity, gastrointestinal obstruction).
7. Expected surgery duration <180 min.
8. Scheduled for urological surgery requiring general anesthesia and laryngeal mask insertion.
9. Voluntary participation with signed informed consent.

Exclusion Criteria:

Baseline measurements: Severe hypertension (SBP >160 mmHg or DBP >100 mmHg), heart rate <60 bpm or >100 bpm.

2. History of long-term alcohol, sedative, or analgesic use; allergy to any study drugs.

3. Severe dysfunction of vital organs (heart, lung, liver, kidney, nervous system), neuromuscular diseases, hyperthyroidism, obstructive sleep apnea syndrome.

4. History of mental disorders or cognitive impairment severe enough to hinder understanding or cooperation with the study.

5. Preoperative administration of sedative-hypnotics (including benzodiazepines and barbiturates).

6. Upper respiratory tract infection within 1 month before surgery. 7. Participation in other clinical studies within the past 3 months. 8. Other conditions deemed unsuitable for the trial by the investigator.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with positive laryngeal mask insertion response | Perioperative
  If the patient has movement during laryngeal mask insertion, twitching at the corner of the mouth, coughing, frowning, tearing, laryngospasm, bispectral index not decreasing to below 60, an increase in heart rate or blood pressure of more than 20% of the baseline value within 2 minutes after laryngeal mask insertion, tachycardia (heart rate >120 beats per minute), or hypertension (systolic blood pressure >180 mmHg), and one of these occurs, it is determined as a positive laryngeal mask insertion reaction; otherwise, it is negative.

SECONDARY OUTCOMES:
Number of adverse reactions | Perioperative
  Blood pressure elevation (systolic blood pressure/diastolic blood pressure >20% baseline), hypotension (systolic blood pressure/diastolic blood pressure <20% baseline or <85/50 mmHg), bradycardia (heart rate <50 bpm), tachycardia (heart rate >100 bpm), hypoxemia (pulse oximetry <92%), When 2 ml of propofol is injected, the patient is asked if there is any injection pain.
Number of successful cases of laryngeal mask placement | Perioperative
  Number of successful cases of laryngeal mask placement
Adverse reactions such as pain, dizziness, headache, nausea and vomiting, sore throat, chills, choking, agitation, hoarseness of voice, and Intraoperative knowledge | Perioperative
  The number of adverse reactions

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-03-19): https://cdn.clinicaltrials.gov/large-docs/15/NCT07096115/Prot_SAP_ICF_000.pdf